CLINICAL TRIAL: NCT07380360
Title: Evaluation of Immediate Implant Placement Accuracy Using a Dynamic Navigation System. "Randomized Clinical Trial"
Brief Title: An Immediate Implant Will be Placed Using the MiniNaviDent System and Static Guide. A Postoperative CBCT Scan Will Then be Acquired and Superimposed Onto the Preoperative CBCT Scan to Assess and Compare Implant Deviation Relative to the Preoperative Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecIM012333
Record Dates: First submitted 2025-12-05; First posted 2026-02-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Remaining Root; Tooth Extraction
Keywords: immediate implant; dynamic navigation; static guide; CBCT superimposition; guided implant surgery

STUDY DESIGN:
Intervention Model Description: All participants will receive immediately placed implants following extraction
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic navigation-guided implant placement (Experimental): Dental implant osteotomy preparation and implant insertion performed using a dynamic navigation system to guide implant placement in real time according to the digital plan (CBCT-based planning with intraoperative navigation guidance)
  Interventions: Device: Dynamic navigation system-assisted dental implant placement
- Static guided implant placement (Active Comparator): Implant placement performed using a patient-specific CAD/CAM static surgical guide fabricated from the digital plan.
  Interventions: Device: CAD/CAM static surgical guide-assisted dental implant placement

INTERVENTIONS:
Device: Dynamic navigation system-assisted dental implant placement — Dental implant placement performed using a dynamic computer-assisted navigation system with real-time guidance. The implant position is planned pre-operatively using CBCT (and intraoral scan data if applicable). During surgery, the system tracks the patient reference and the drill/handpiece and displays real-time guidance to follow the planned implant trajectory for osteotomy preparation and implant insertion.
  Device name: mini Navident
  Arms: Dynamic navigation-guided implant placement
Device: CAD/CAM static surgical guide-assisted dental implant placement — Dental implant placement performed using a patient-specific CAD/CAM static surgical guide. The guide is designed from the digital implant plan (CBCT and, if applicable, intraoral scan) and fabricated (e.g., 3D printed). The static guide (with sleeves) is used to guide osteotomy preparation and implant insertion according to the planned implant position.
  Arms: Static guided implant placement

SUMMARY:
This clinical study aims to evaluate implant deviation during immediate implant placement using dynamic navigation. By utilizing implant planning software, two CBCT scans (preoperative and postoperative) will be superimposed to assess the accuracy of dynamic navigation in immediate implant placement, which is considered a more complex procedure compared to delayed implant placement

DETAILED DESCRIPTION:
First, a fiducial marker will be placed in the patient's mouth, followed by a CBCT scan with the marker in position. The implant will then be virtually planned using implant planning software. Using the MiniNaviDent system and the fiducial marker, the implant will be placed. After placement, a postoperative CBCT scan will be obtained. The postoperative scan will be superimposed onto the preoperative scan to measure implant deviation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients at least 21 years old.
2. Systemically healthy patients with no effect on the surgery.
3. At least one hopeless maxillary or mandibular tooth to be restored using an implant.
4. At least six residual teeth in the affected jaw.

Exclusion Criteria:

1. A medical condition or medication that would impair bone healing.
2. Poor oral hygiene
3. Alcohol users.
4. Smoking more than 10 cigarettes per day.
5. History of head and neck radiotherapy.
6. Pregnant females.
7. Uncontrolled hypertensive or diabetic patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Coronal deviation (mm) Apical deviation (mm) | Pre-op CBCT and post-op CBCT within 7 days after surgery
  Implant deviation was defined as the discrepancy between the planned implant position (as established in the preoperative planning software) and the actual implant position placed using dynamic navigation and a static surgical guide. To quantify this deviation, the postoperative CBCT was superimposed (registered) onto the preoperative planned CBCT, and the resulting spatial differences between the planned and placed implants were measured and reported in millimeters (mm)
Angular deviation (degrees) | Pre-op CBCT and post-op CBCT within 7 days after surgery
  Implant deviation was defined as the discrepancy between the planned implant position (as established in the preoperative planning software) and the actual implant position placed using dynamic navigation and a static surgical guide. To quantify this deviation, the postoperative CBCT was superimposed (registered) onto the preoperative planned CBCT, and the resulting spatial differences between the planned and placed implants were measured and reported in and the angular deviation in degrees was measured.

SECONDARY OUTCOMES:
Total surgical time (minutes) | Intraoperative (day of surgery)
  Total operative time recorded in minutes from first mucosal incision to completion of final implant insertion (last implant fully seated). Time will be recorded by an independent observer using a stopwatch and compared between the dynamic navigation and Static Guide groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided